CLINICAL TRIAL: NCT00883701
Title: Granzymes and Perforin at the Onset of COPD Exacerbations
Brief Title: Granzymes and Perforin at the Onset of Chronic Obstructive Pulmonary Disease (COPD) Exacerbations
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Stelios Lazarou, University of Thessaly
Other Study IDs: SL19021970DM
Record Dates: First submitted 2009-04-16; First posted 2009-04-20 (Estimated); Last update posted 2010-04-29 (Estimated); Status verified 2009-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; exacerbations; perforin; granzymes
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — sputum cells and supernatant
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- COPD patients: COPD patients who undergo exacerbation
- Non COPD patients (controls): Subjects who undergo respiratory infection (acute bronchitis) without COPD or other respiratory illness

SUMMARY:
COPD exacerbations are characterized by an excessive accumulation and activation of inflammatory cells in the airways. It is not known whether this phenomenon represents a risk for for lung damage via the release in the extracellular environment of potent cytolitic cellular granular contents such as granzymes and perforin.

The investigators assess the intracellular expression of granzymes and perforin in neutrophils and large granular lymphocytes (LGL) at the onset of exacerbations compared to stable disease.

The investigators hypothesize that a greater release of intracellular perforin and granzymes from neutrophils and LGL into the extracellular environment occur at exacerbations compared to stable condition and that these changes are more pronounced in COPD patients than in subjects without COPD who undergo respiratory infection.

DETAILED DESCRIPTION:
The course of Chronic Obstructive Pulmonary Disease (COPD) is characterized by exacerbations which lead to significant clinical deterioration and morbidity.COPD exacerbations are characterized by an augmentation of the inflammation that is observed in the airways in stable condition, particularly by excessive accumulation of polymorphonuclear neutrophils and activation of lymphocytes.

It has been suggested that this abnormal increase of inflammatory cells in the airways of COPD patients during exacerbations, might represent a significant risk for excessive proteolytic activity in the airways via the release of their granule contents into the extracellular environment. Large granular lymphocytes (LGL) which include NK and cytotoxic T- cells and neutrophils contain cytolytic molecules such as, granzymes and perforin. Therefore, the inflammatory process during exacerbations might be potentially toxic to the lung. Notably, it was showed that sputum T-lymphocytes (CD8+) from patients with stable COPD express more perforin and are more cytotoxic compared to normal subjects.

However, few previous investigations questioned the role of these cytolytic molecules in the pathophysiology of COPD. Moreover, despite the considerable progress that has been made in understanding the underlying mechanisms in COPD, there have been no studies investigating the expression of perforin or granzymes during COPD exacerbations.

In the present prospective investigation we assess the intracellular expression of granzymes and perforin in neutrophils and LGL cells at the onset of sputum of COPD patients by using flow cytometry.

Subjects and protocol:

COPD subjects will be examined at the onset of an exacerbation and in stable condition. The definition of an exacerbation will be based on the criteria described by Anthonisen, requiring either the presence of at least two major symptoms (increase in dyspnea, sputum production, purulence) or of one major symptom in addition to at least one minor (wheeze, cough, nasal discharge, sore throat, fever), for two consecutive days.

In addition we will assess the expression of granzymes and perforin in neutrophils and LGL cells of subjects without COPD(controls) who will be recruited by consecutive sampling among those subjects who seek medical assistance at the clinic during the study period and they satisfy all the following criteria: i) absence of COPD, Asthma, pneumonia, evidence of lung cancer, bronchiectasis, interstitial lung disease or other respiratory disease ii) initiation of symptoms diagnostic for respiratory infection in the past 72 hours, iii) abstention from any new therapeutic intervention, and iv) absence of any signs suggestive of condition requiring hospitalization. Control subjects will be examined at the onset of respiratory infections and at stable condition. The definition of a respiratory infection require the presence of one of the following symptoms such as dyspnea, sputum production, purulence, cough, ± fever, for two consecutive days. Stable condition for controls will be defined as absence of respiratory infection/exacerbation based on symptoms.

The study is approved by the Research Ethics Committee of the Hospital . Sputum induction and processing Sputum will be induced at exacerbation or respiratory infection and in stable condition (at least 8 weeks after exacerbation) of the same patient and control subject respectively; samples will be processed for analysis of inflammatory cells and cytokines and microbiology. Sputum will be induced via inhalation of a hypertonic saline solution aerosol (Ultraneb 2000; DeVilbiss; Somerset, PA).

Antibody labeling:

The following mouse anti-human monoclonal antibodies will be used for labeling sputum cells: phycoerythrin-conjugated antiCD3 (PE-CD3), phycoerythrin-5-conjugated (antiCD4-PCy5), fluorescein isothiocyanate-conjugated anti-perforin-antibody, (antiperforin-FITC) and fluorescein isothiocyanate-conjugate will be also used for competitive detection of intracellular perforin and granzymes. The "a intraprep kit" (Beckman-Coulter Inc Fullerton Ca, USA). Isotyping antibodies mouse antimouse IgG will be used as controls (Immunotech; Marseille, France). For labeling cell surface antigens 1x106 cells in suspension will be incubated with normal bovine serum to block the unspecific binding (blocking reagent), and then the monoclonal antibody/ antibodies will be added in excess (according to manufacturer's instruction) for 45 min at 10°C in the dark and washed three times with PBS plus 10% FCS. For intracellular perforin and granzymes staining, cells will be subsequently incubated in a permeabilization reagent (Intraprep; Beckman Coulter; Fullerton, CA) for 10 min. As a control, unlabeled antiperforin (or antigranzyme) at molar excess will be used after permeabilization and then antiperforin (or antigranzyme) FITC will be added without washing and incubated for 30 min at room temperature (competitive labeling). After staining, the samples will be washed with PBS plus 10% FCS and will be immediately analyzed using flow cytometry.

Flow Cytometric analysis:

The sputum samples prepared as described above will be analyzed on a fluorescence activated cytometer (EPICS ELITE; Coultronics; Louton, UK). Cells will be tightly gated by volume and complexity on a forward (0o) and side-light scattering (90o) mode. At least 105 cells were analyzed in each session. PCy-5-conjugated anti-human CD45 monoclonal antibodies (Dako; Ely, UK) will be used as pan-leukocyte stain to exclude non leukocyte events by logical gating. The percentage of one-color, two-color, and three-color positive cells will be measured and the mean channel value as well as the relative fluorescence intensity (RFI) corresponding to the antigen density will be estimated. The QC-Combo Kit (FCSC; San Jun, Puerto Rico) will be used for quantification of antibody binding and day-to-day instrument calibration (amplification and compensation settings of the flow cytometer) will be routinely carried out. Gating will be performed according to forward and side scattering and CD45 expression. Positive cells within the neutrophilic and lymphocytic population will be measured as percentages of each cell population.

Following the above methodology we will asses the expression of perforin in neutrophils and LGL cells and the expression of granzymes in neutrophils and LGL cells both in exacerbation and in stable COPD.

ELIGIBILITY:
COPD patients

Inclusion Criteria:

* All COPD patients who seek medical assistance at the clinic during the study period will be asked about COPD exacerbation related symptoms-medical history and then they will be included in the study if they satisfied all the following criteria:

  * COPD diagnosis according to the GOLD Consensus Statement
  * initiation of symptoms diagnostic for COPD exacerbation in the past 72 hours
  * abstention from any new therapeutic intervention
  * absence of any signs suggestive of severe exacerbation requiring hospitalization

Control subjects

Inclusion Criteria:

* Subjects who seek medical assistance at respiratory clinic for symptoms suggesting acute bronchitis (dyspnea, sputum production, purulence, wheeze, cough)

  * medical history free of COPD, Asthma, pneumonia, other chronic respiratory disease or congestive cardiac failure,
  * initiation of symptoms in the past 72 hours,
  * abstention from any new therapeutic intervention, and
  * absence of any signs suggestive of clinical condition requiring hospitalization.

Exclusion Criteria:

* Patients with Asthma or other respiratory disease will be excluded from this study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients
  Subjects are recruited from a community based outpatient primary medical clinic by consecutive sampling.
  Control subjects
  Subjects who seek medical assistance for symptoms suggesting acute bronchitis (dyspnea, sputum production, purulence, wheeze, cough) are recruited from a community based outpatient primary medical clinic by consecutive sampling.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2002-12; Primary Completion 2008-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Expression of granzymes and perforin in neutrophiles and LGL sputum cells | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Demos Makris, MD, Study Director — University of Thessaly
Locations (1):
- University Hospital Larisa, Larissa, Thessaly, Greece